CLINICAL TRIAL: NCT03509766
Title: Randomized Evaluation of Ten Allergy Skin Prick Test Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: NA_00092406
Record Dates: First submitted 2013-12-27; First posted 2018-04-26 (Actual); Results first posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Allergic Rhinitis; Asthma; Food Allergy; Skin Testing
Keywords: allergic; rhinitis; allergy; asthma; food allergy; skin testing; skin prick test
MeSH Terms: conditions — Rhinitis, Allergic; Asthma; Food Hypersensitivity; Rhinitis; Hypersensitivity | interventions — Skin Tests

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Neither the subject nor the technician are masked as to which device is being placed. However, the investigator who reads the skin prick test results is blinded as to which device is which.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Skin testing (Experimental): All subject both allergic and non-allergic will be tested. There is only one (1) arm.
  Interventions: Device: Histamine skin testing

INTERVENTIONS:
Device: Histamine skin testing — skin testing using histamine
  Other Names: skin test device; skin prick test device

SUMMARY:
The goal of this study is to compare ten current and readily available FDA approved allergy skin prick devices to determine the most sensitive and specific product and methods used for the diagnosis of allergic disease. The primary outcome will be to determine the analytical sensitivity and specificity of all ten skin prick devices by measuring wheal and flare response to histamine and control diluent in 1mm increments. Secondary outcomes include comparison of skin prick technique, optimum histamine concentration, patient comfort, reproducibility, and the comparability of high-resolution digital images.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 with or without allergic disease

Exclusion Criteria:

* severe concurrent illness
* uncontrolled asthma
* extensive eczema
* urticaria
* dermatographism
* pregnancy
* those taking antihistamines within the previous 10 days
* topical steroids
* immunomodulatory drugs
* long term use of oral steroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- John Hopkins Asthma and Allergy Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Skin Testing: All subjects both allergic and non-allergic will be tested. There is only one (1) arm.
  Histamine skin testing: skin testing using histamine
Period: Overall Study
Arm/Group | Skin Testing
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Skin Testing
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 6
  Female | 18

OUTCOME MEASURES:

1. Primary Outcome: Wheal Response
Description: Compare Wheal response among devices using 1mm precision. SPT test will be read at 15 min time point. The maximum wheal diameter will be recorded for each of ten skin prick devices. 3mm (and 2mm above negative control) qualify as a positive test.
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Skin Testing
Number analyzed (Participants) | 24
mm | 6.8 (0.4)

2. Primary Outcome: Sensitivity
Description: Sensitivity is calculated by dividing the true positive wheals divided by true positives plus false negatives and multiplying by 100. For example one false negative out of 24 tests equals a sensitivity of 95.8%.
Time Frame: 15 minutes
Measure: Number; unit: percentage of tests true positive
Arm/Group | Skin Testing
Number analyzed (Participants) | 24
percentage of tests true positive | 95.8

3. Secondary Outcome: Skin Prick Techniques/Methodology Ratio
Description: Compare 1mg/ml versus 6mg/ml histamine base for Duotip II twist method. Maximum wheal diameter is measured for each concentration.
Time Frame: 15 minutes
Population: All 24 subjects received DuoTip II with both 1mg/ml and 6mg/ml histamine. This 24 vs 24 SPT in 24 total subjects.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- 1 Versus 6mg: 1 versus 6mg histamine
Arm/Group | 1 Versus 6mg
Number analyzed (Participants) | 24
ratio | 1 (.01)

ADVERSE EVENTS:
Groups:
- Adverse Events: no adverse events or reactions were reported. Events were recorded during the procedure and for 30 days following the procedure. Both serious and and non life threatening adverse vents were recorded.
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No